CLINICAL TRIAL: NCT02034591
Title: Bioavailability of Apixaban Oral Solution Administered Through a Nasogastric Tube in the Presence of Boost® Plus and Apixaban Administered as Crushed Tablet Through a Nasogastric Tube Relative to Apixaban Oral Solution in Healthy Subjects
Brief Title: Phase 1 Oral Solution and Crushed Tablet Relative Bioavailability Study of Apixaban When Administered Through a Nasogastric Tube in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-111
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A-Apixaban (Experimental): Solution Apixaban 5 mg ( 0.4 mg/ml oral solution x 12.5 ml) through mouth or oral syringe
  Interventions: Drug: Apixaban
- Arm B-Apixaban (Experimental): Oral Solution Apixaban 5 mg single dose (0.4 mg/mL oral solution x 12.5 mL) after 180 mL of Boost Plus®, followed by 60 mL of Boost Plus® via same NGT
  Interventions: Drug: Apixaban; Dietary Supplement: Boost Plus
- Arm C-Apixaban (Experimental): Single dose crushed Apixaban tablet 5 mg (5 mg tablet crushed and suspended in 60 mL Dextrose 5% in water (D5W)) through NGT
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS-562247
Dietary Supplement: Boost Plus
  Arms: Arm B-Apixaban

SUMMARY:
The purpose of this study is to assess the bioavailability of Apixaban oral solution administered through an Nasogastric Tube (NGT) in the presence of Boost® Plus and Apixaban administered as crushed tablet through a nasogastric tube relative to Apixaban solution administered orally in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Any history or evidence of abnormal bleeding or coagulation disorders, intracranial hemorrhage, or abnormal bleeding (including heavy menstrual bleeding that has resulted in anemia within the past 1 year) or coagulation disorders in a first degree relative

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries, LLC D/B/A Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- [Derived] Song Y, Wang X, Perlstein I, Wang J, Badawy S, Frost C, LaCreta F. Relative Bioavailability of Apixaban Solution or Crushed Tablet Formulations Administered by Mouth or Nasogastric Tube in Healthy Subjects. Clin Ther. 2015 Aug;37(8):1703-12. doi: 10.1016/j.clinthera.2015.05.497. Epub 2015 Jul 15. PMID 26188837
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants were enrolled; 21 were randomized and treated. Reasons for non-randomization include 11 no longer met study criteria, 1 withdrew consent and 4 for other, not specified reasons. 20 participants completed the study; 1 withdrew consent on day 4 of treatment.
Groups:
- Treatment A, Then Treatment B, Then Treatment C; Treatment A, Then Treatment C, Then Treatment B; Treatment B, Then Treatment A, Then Treatment C; Treatment B, Then Treatment C, Then Treatment A; Treatment C, Then Treatment A, Then Treatment B; Treatment C, Then Treatment B, Then Treatment A: Each participant was given three interventions, one per period, with a 4 day washout in between periods
  Treatment A: Single dose apixaban 5 milligrams (mg) oral solution (OS) (0.4 milligrams per milliliter (mg/mL) x 12.5 milliliters (mL) administered by mouth via oral syringe
  Treatment B: Single dose apixaban 5 mg OS (0.4 mg/mL x 12.5 mL) administered via nasogastric tube (NGT) after 180 mL of Boost® Plus, followed by 60 mL of Boost® Plus via same NGT
  Treatment C: Single dose apixaban 5 mg (5 mg tablet crushed and suspended in 60 mL 5% dextrose in water (D5W) administered via NGT
Period: Overall Study
Arm/Group | Treatment A, Then Treatment B, Then Treatment C | Treatment A, Then Treatment C, Then Treatment B | Treatment B, Then Treatment A, Then Treatment C | Treatment B, Then Treatment C, Then Treatment A | Treatment C, Then Treatment A, Then Treatment B | Treatment C, Then Treatment B, Then Treatment A
Started | 4 | 3 | 4 | 3 | 4 | 3
Completed | 4 | 3 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- All Treatment Groups: All Randomized Participants
Arm/Group | All Treatment Groups
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 36.7 [22 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean of the Maximum Observed Plasma Concentration (Cmax) of Apixaban
Description: Maximum observed plasma concentration (Cmax) is measured in nanograms per milliliter (ng/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available pharmacokinetic (PK) data
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Treatment A: Single dose apixaban 5 milligrams (mg) oral solution (OS) (0.4 milligrams per milliliter (mg/mL) x 12.5 milliliters (mL) administered by mouth via oral syringe
- Treatment B: Single dose apixaban 5 mg OS (0.4 mg/mL x 12.5 mL) administered via nasogastric tube (NGT) after 180 mL of Boost® Plus, followed by 60 mL of Boost® Plus via same NGT
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 20 | 20
ng/mL | 179.116 [164.855 to 194.611] | 122.145 [112.011 to 133.196]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.682, 90% CI 2-sided [0.621 to 0.748]

2. Primary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero Extrapolated to Infinite Time AUC(INF) of Apixaban
Description: AUC(INF) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available PK data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 20 | 20
ng*h/mL | 1397.666 [1330.658 to 1468.049] | 1136.380 [1065.716 to 1211.729]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.813, 90% CI 2-sided [0.766 to 0.863]

3. Primary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Apixaban
Description: AUC(0-T) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available PK data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 20 | 20
ng*h/mL | 1372.836 [1306.240 to 1442.828] | 1112.493 [1041.751 to 1188.038]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.810, 90% CI 2-sided [0.764 to 0.860]

4. Secondary Outcome: Adjusted Geometric Mean of the Maximum Observed Plasma Concentration (Cmax) of Apixaban
Description: Maximum observed plasma concentration (Cmax) is measured in nanograms per milliliter (ng/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available PK data
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Treatment C: Single dose apixaban 5 mg (5 mg tablet crushed and suspended in 60 mL 5% dextrose in water (D5W) administered via NGT
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 20 | 21
ng/mL | 179.116 [164.855 to 194.611] | 158.371 [145.849 to 171.968]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.884, 90% CI 2-sided [0.830 to 0.942]

5. Secondary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time [AUC(INF)] of Apixaban
Description: AUC(INF) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available PK data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 20 | 21
ng*h/mL | 1397.666 [1330.658 to 1468.049] | 1327.248 [1246.871 to 1412.806]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority or Other; Ratio of Adjusted Geometric Means = 0.950, 90% CI 2-sided [0.905 to 0.997]

6. Secondary Outcome: Adjusted Geometric Mean of the Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] of Apixaban
Description: AUC(0-T) is measured in nanogram hours per milliliter (ng*h/mL)
Time Frame: Pre-dose and 0.25, 0.50, 1, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 60, 72 hours post-dose for each intervention
Population: All randomized participants with available PK data
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 20 | 21
ng*h/mL | 1372.836 [1306.240 to 1442.828] | 1300.728 [1220.374 to 1386.374]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.947, 90% CI 2-sided [0.903 to 0.994]

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths or Discontinuation of Study Drug Due to AEs
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during the study and up to 28 days past study discontinuation. The select AEs were determined using the Medical Dictionary for Regulatory Activities (MedDRA, v15.1) and graded using the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0
Time Frame: Day 1 to 30 days after last dose of study drug
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 20 | 21
participants
  SAE | 0 | 0 | 1
  Treatment-Related AE | 0 | 1 | 1
  Deaths | 0 | 0 | 0
  Treatment-Related Deaths | 0 | 0 | 0
  Discontinuation of Study Drug Due to AEs | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Marked laboratory abnormalities were defined as laboratory assessments meeting the following investigator-specified criteria: Leukocytes >1.2* upper limits of normal (ULN) , Basophils >3%, Eosinophils >1.5*ULN, Blood Urine >=2, Red Blood Cell (RBC) Urine >=2, White Blood Cell (WBC) Urine >=2
Time Frame: Day 1 to 30 days after last dose of study drug
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 20 | 21
participants
  Leukocytes | 0 | 1 | 0
  Basophils | 1 | 0 | 0
  Eosinophils | 0 | 1 | 0
  Blood, Urine | 1 | 1 | 0
  RBC, Urine | 0 | 2 | 1
  WBC, Urine | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to 30 days after last dose of study drug
Arm/Group | Treatment A | Treatment B | Treatment C
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/21
Other Adverse Events (participants affected / at risk) | 6/20 | 3/20 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=20) | Treatment B (N=20) | Treatment C (N=21)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=20) | Treatment B (N=20) | Treatment C (N=21)
Haematoma (Vascular disorders) | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less